CLINICAL TRIAL: NCT00000319
Title: Buprenorphine Maintenance Dose Schedule and Treatment Setting
Brief Title: Buprenorphine Maintenance Dose Schedule and Treatment Setting - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-09803-2; R01DA009803 (NIH); R01-09803-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the efficacy of treating opioid-dependent individuals with buprenorphine on a thrice-weekly schedule compared to daily dosing.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-06; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Depression
Withdrawal symptoms
Opioid and cocaine use
Social and psychological functioning
AIDS risk behavior
Opiate withdrawal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Yale University
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States